CLINICAL TRIAL: NCT02354911
Title: A Randomized, Double-Blind, Placebo-Controlled, Cross-Over Study of the Safety and Efficacy of Autologous Immunoregulatory Dendritic Cells in Patients With Type 1 Diabetes
Brief Title: Autologous Immunoregulatory Dendritic Cells for Type 1 Diabetes Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding for study not procured.
Sponsor: DiaVacs, Inc. (Industry)
Collaborators: West Penn Allegheny Health System (Other); University of Pittsburgh Medical Center (Other); Stanford University (Other); University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DV-0100-101
Record Dates: First submitted 2015-01-27; First posted 2015-02-03 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Type 1 Diabetes
Keywords: Immunomodulation
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immunoregulatory Dendritic Cells (iDC) (Experimental): Biological intervention consisting of autologous dendritic cells treated in vitro to convert to active immunoregulatory dendritic cells.
  Interventions: Biological: Immunoregulatory Dendritic Cells
- Placebo Control (Placebo Comparator): Saline injections administered blinded to subject and all study staff except for research pharmacist who is not involved in study conduct
  Interventions: Other: Placebo Comparator: Placebo Control

INTERVENTIONS:
Biological: Immunoregulatory Dendritic Cells — Autologous dendritic cells harvested by leukapheresis and engineered ex vivo via incubation with antisense DNA oligonucleotides targeting the primary transcripts of CD40, CD80 and CD86. The ex vivo engineered product is then administered via blinded intradermal injection in the peri-umbilical region of the abdomen given as 4 separate injections at 2-week intervals (~10 million cells/injection).
  Other Names: iDC
  Arms: Immunoregulatory Dendritic Cells (iDC)
Other: Placebo Comparator: Placebo Control — Blinded intradermal injections in the peri-umbical region of the abdomen given as 4 separate injections at 2-week intervals
  Arms: Placebo Control

SUMMARY:
The purpose of this study is to determine whether dendritic cells collected via leukapheresis and incubated with antisense DNA oligonucleotides and then injected back into the same subject will serve as modulators of the immune system in a manner that disrupts the autoimmune process responsible for the destruction of pancreatic beta cells in subjects with new onset type 1 diabetes.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled cross study designed to evaluate the safety and efficacy of autologous immunoregulatory dendritic cells (iDC) in patients with type 1 diabetes. To do this, a total of 24 subjects with recent onset (<100 days from diagnosis) type 1 diabetes will have circulating dendritic cells harvested via leukapheresis. The harvested dendritic cells will then be incubated in vitro with antisense DNA oligonucleotides targeting the primary transcripts of cluster of differentiation antigen 40 (CD40), cluster of differentiation antigen 80 (CD80) and cluster of differentiation antigen 86 (CD86). These engineered dendritic cells will then be given as autologous intradermal injections (4 injections administered at 2 week intervals) in the subject' peri-umbilical region. The hypothesis is that the injected cells will generate immunoregulatory cells that suppress the autoimmune process responsible for the development of type 1 diabetes via destruction of the subject's pancreatic beta cells.

Employing a cross-over design, all subjects will undergo leukapheresis at the outset. Twelve subjects will be randomly assigned to receive cell injections at the outset while the other 12 subjects will receive sham injections and serve as controls. At the end of 12 months, all subjects will cross-over to the alternative treatment and continue to be followed for an additional 12 months. (Note: The subjects assigned to receive the cell therapy for this segment will receive injections of their autologous cells harvested and engineered at the time of the leukapheresis performed at study entry. The engineered cells will be stored frozen until needed for administration. This design will test whether treatment later (>1 year after diagnosis) is as effective as immediate treatment (<100 days from the diagnosis of type 1 diabetes).

As an added safety measure, the first 6 subjects randomized will all be over the age of 18. When the last of these 6 subjects complete 3 months of observation following the initiation of therapy, the age for enrollment will be lowered to age 16 for the next 6 subjects unless safety observations dictate otherwise. When all subjects in this cohort have been enrolled, the age for enrollment will be lowered to age 14 unless advised otherwise by the independent Data Safety Monitoring Board. When all subjects in this cohort have completed observation for 3 months, the age for enrollment will be lowered to age 12 following clearance by the Data Safety Monitoring Board.

If this therapy is successful, the subjects' remaining beta cell mass will be preserved and hopefully expanded once the autoimmune process is slowed or stopped. This outcome will be assessed indirectly using plasma c-peptide concentrations following ingestion of a standardized mixed meal at the end of 12 and 24 months of therapy. If the treatment is successful, glucose control should improve and be detectable via measurement of hemoglobin A1c (measure of long-term control), fasting plasma glucose concentrations and the plasma glucose concentrations following ingestion of the standardized mixed meal. In addition, the total daily insulin requirements should decrease. These measures of glucose control will be assessed at baseline and then at 3, 6, 9, 12, 15, 18, 21 and 24 months.

Immune markers will also be profiled at 3 month intervals to assess potential tolerogenic effects of the therapy. To this end, numbers of potentially tolerogenic/regulatory T-cells, B-cells and dendritic cells in the circulating peripheral blood monocyte population will be assessed. In addition, analysis of selected populations of T-cells, B-cells and dendritic cells will be conducted over the entire study period in an attempt to identify molecular signatures correlated with the clinical response.

Finally, in addition to the routine safety laboratory measurements, all reported adverse events will be examined in detail to characterize the safety aspects of the therapy. The review of these safety data will be guided by an independent Data Safety Monitoring Board which will meet at least semi-annually to review the accrued data.

ELIGIBILITY:
Inclusion Criteria:

1. Fully executed, Institutional Review Board (IRB) approved, informed consent form
2. New onset type 1 diabetes randomized within 100 days of diagnosis
3. Positive for at least one islet cell auto-antibody; GAD, insulin (if sample within 7 days of the onset of insulin therapy), islet antibody 2 (IA-2), zinc transporter 8 antibody (ZnT8), and/or islet cell antibody (ICA)
4. Peak plasma c-peptide concentration >0.2 pmol/mL after ingestion of a standardized mixed meal
5. Serologic evidence of prior Epstein-Barr virus (EBV) infection
6. Immunoreactivity to alloantigens in mixed leukocyte culture and reactivity to viral antigens (CEF Pool Assay) in vitro
7. Adequate peripheral venous access for leukapheresis
8. Female participants with childbearing potential must agree to use effective birth control during study participation. Reliable and effective forms of birth control include: true abstinence, intrauterine device (IUD), hormonal-based contraception, double-barrier contraception (condom or occlusive cap (diaphragm or cervical cap) + spermicide, or surgical sterilization (vasectomy for male partner, tubal ligation or hysterectomy).
9. Sexually active male participants must agree to use condoms during intercourse

Exclusion Criteria:

1. History of enrollment in a drug, or biologic therapy clinical trial within past 12 months impacting the immune system
2. Prior or current therapy known to cause a significant, ongoing change in the course of type 1 diabetes or immune status
3. Evidence of active infection at screening (e.g. "common cold", influenza, hepatitis, tuberculosis, EBV, cytomegalovirus (CMV), herpes simplex virus (HSV), HIV, varicella, chlamydia, evidence of serious fungal infection) or screening laboratory evidence consistent with active microbial, viral, or fungal infection (minor cutaneous fungal infection is not an exclusion)
4. Leukopenia (<3,000 leukocytes/microliter, neutropenia (<1,500 neutrophils/microliter), lymphopenia (<800 lymphocytes/microliter) or thrombocytopenia (<125,000 platelets/microliter)
5. Positive screen for HIV, tuberculosis, hepatitis B, hepatitis C, herpes simplex virus 1 (HSV1) or herpes simplex virus 2 (HSV2) infection
6. Vaccination with any live vaccine product within the 3 months prior to the first cycle of study agent administration
7. Female subjects pregnant or unwilling to defer pregnancy for the study period
8. Females lactating at screening
9. History of significant heart disease (e.g., myocardial infarction, coronary artery disease, angina pectoris, arrhythmia, uncontrolled hypertension, congestive heart failure, structural defects)
10. Liver disease with alanine transaminase (ALT) or aspartate aminotransferase (AST) >3 times the upper limit of normal
11. Impaired renal function with a serum creatinine concentration > 1.5.
12. Any other significant immune disorder including, but not limited to, rheumatoid arthritis, systemic lupus erythematous, multiple sclerosis, vitiligo, ankylosing spondylitis and celiac disease. (Thyroiditis treated with a stable dose of thyroid replacement therapy is allowed.)
13. Any condition that interferes with accurate measurement of glycated hemoglobin (hemoglobin A1C)
14. Any condition that, in the investigator's opinion, may compromise continuous study participation or confound study results
15. Any planned vaccinations scheduled prior to end of study participation
16. Chronic treatment with systemic corticosteroids (topical or inhaled corticosteroids are allowed)
17. Current use of diabetes medications other than insulin
18. Anticipated need for any of the following therapies during the 24-month study period:

    * Radiation therapy
    * Oncologic chemotherapy
    * Corticosteroids except for very short courses (≤ 2 weeks)
    * Agents used to treat attention deficit and hyperactivity disorder (ADHD)
    * Any protein, particle or cell vaccine immunomodulation therapy

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the mean 2-hour area under the curve (AUC) for plasma c-peptide at 12 and 24 months | 12 and 24 months
  Mean 2-hour area under the time-concentration curve for plasma c-peptide following ingestion of a standardized mixed meal compared across treatment groups at end of Segment 1 (12 months) and Segment 2 (24 months)

SECONDARY OUTCOMES:
Reported adverse events | 12 months; 12 to 24 months and 0 to 24 months
  All reported adverse events for treatment compared to placebo control group across each treatment period
Change from baseline in number of potentially-tolerogenic/regulatory T-cells, B-cells and dendritic cells in circulating peripheral blood mononuclear cell fraction | 3,6,9,12,15,18,21 and 24 months
  Numbers of potentially-tolerogenic/regulatory T-cells, B-cells and dendritic cells in circulating peripheral blood mononuclear cell fraction assessed at 3 month intervals over the course of both treatment periods based on defined cell markers
Change from baseline in sub-populations of T-cells | 3,6,9,12,15,18,21 and 24 months
  Sub-populations of T-cells in iDC treatment group compared to placebo group assessed at 3 month intervals throughout the course of both segments of the trial
Change from baseline in sub-populations of B-cells | 3,6,9,12,15,18,21 and 24 months
  Sub-populations of B-cells in iDC treatment group compared to placebo group assessed at 3 month intervals throughout the course of both segments of the trial
Change from baseline in sub-populations of dendritic cells | 3,6,9,12,15,18,21 and 24 months
  Sub-populations of dendritic cells in iDC treatment group compared to placebo group assessed at 3 month intervals throughout the course of both segments of the trial
Change from baseline in Fasting Plasma Glucose | 3, 6, 9, 12,15,18,21, and 24 months
  Plasma glucose concentration following an overnight fast of at least 8 hours duration
Change from baseline in Hemoglobin A1c | 3, 6, 9, 12,15,18,21, and 24 months
  Measurement of hemoglobin A1c is the well-established measure of glucose control reflecting the "integrated" glycemic exposure over the past 90 to 120 days
Change from baseline in the baseline corrected, 2-hour AUC for glucose at 12 and 24 months | 12 and 24 months
  Baseline corrected, 2-hour AUC for plasma glucose following ingestion of a standardized mixed meal
Change from baseline in Total Daily Insulin Dose | 3, 6, 9, 12,15,18,21, and 24 months
  The cumulative total daily insulin dose collected as the average for the 3-day period immediately prior to the respective clinic visits. This includes all forms of insulin used by the subject

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Trucco, PhD, Study Chair — Institue of Cellular Therapeutics, Allegheny General Hospital, Pittsburgh, PA

REFERENCES:
- [Derived] Phillips BE, Garciafigueroa Y, Engman C, Trucco M, Giannoukakis N. Tolerogenic Dendritic Cells and T-Regulatory Cells at the Clinical Trials Crossroad for the Treatment of Autoimmune Disease; Emphasis on Type 1 Diabetes Therapy. Front Immunol. 2019 Feb 6;10:148. doi: 10.3389/fimmu.2019.00148. eCollection 2019. PMID 30787930